CLINICAL TRIAL: NCT05456503
Title: Imaging Tau Accumulation in FTLD and Atypical Alzheimer's Disease Using the PET Ligand [18F]-PI-2620
Brief Title: PET Imaging Tau Accumulation in FTLD and Atypical Alzheimer's Using [18F]-PI-2620
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 849866
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Frontotemporal Lobar Degeneration; Alzheimer Disease; Cognitively Normal
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Alzheimer Disease | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cognitively and neurologically normal adults (CN) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Non-amnestic Alzheimer's Disease (AD) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Frontotemporal lobar degeneration from tauopathy (FLTD-tau) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Frontotemporal lobar degeneration from TDP-43 (FLTD-TDP) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Frontotemporal lobar degeneration from mutation in the MAPT gene (genetic FLTD-tau) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Frontotemporal lobar degeneration from mutation in the GRN gene or frame 72 of chromosome 9 (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620
- Amnestic Mild Cognitive Impairment Alzheimer's Disease (MCI/aAD) (Experimental): One PET imaging scan using the [18F]-PI-2620 tracer
  Interventions: Drug: [18F]-PI-2620

INTERVENTIONS:
Drug: [18F]-PI-2620 — Radiotracer

SUMMARY:
The investigators will compare [18F]-PI-2620 tau PET scans from patients with frontotemporal lobar degeneration (FTLD), patients with non-amnestic presentations of Alzheimer's disease (naAD), and demographically matched cognitively normal subjects.

DETAILED DESCRIPTION:
The current study is a companion imaging study to IRB# 842873, "University of Pennsylvania Centralized Observational Research Repository on Neurodegenerative Disease" (UNICORN). All participants in the current study must be concurrently enrolled in UNICORN. UNICORN is an observational study that aims to collect and store cross-sectional and longitudinal data from brain imaging, clinical and neuropsychological assessment, biomarker assays, and genetic testing of participants to improve clinical assessment and basic scientific understanding of multiple neurodegenerative conditions. The UNICORN cohort includes neurodegenerative disease patients who have been evaluated by trained neurologists in the Penn Cognitive Neurology Clinic according to published clinical research diagnostic criteria and reviewed at a weekly multidisciplinary consensus conference; as well as individuals with normal cognition recruited from the general community or from among caregivers/relatives of patients participating in research. As part of the UNICORN study, participants are asked to undergo periodic (typically annual) magnetic resonance imaging (MRI) and clinical/neuropsychological assessment. All participants' biological samples may be subjected to research genetic testing analyses. Results from these analyses are considered research, and as such are used for research purposes only. UNICORN participants are also asked to undergo a one-time lumbar puncture to assess cerebrospinal fluid protein levels, including amyloid-ß1-42, an established biomarker for Alzheimer's disease (AD) neuropathologic change. As an alternative method of assessing amyloid status, some UNICORN participants may have previously undergone an [18F] florbetaben amyloid PET scan under protocol #824869. The procedure for detecting amyloid could also be a lumbar puncture that was performed for clinical purposes or an amyloid PET scan, performed either clinically or for research purposes.

Participants will be screened according to the study selection criteria, based on self-report, information provided by caregivers, and medical history available through PennChart or through the Integrative Neurodegenerative Disease Database (INDD). All screening/enrollment documentation will come from the parent study, IRB# 842873 UNICORN. Participants will provide written informed consent for this protocol before beginning any study specific procedures. Participants must satisfy all eligibility criteria and consent to [18F]-PI-2620 PET imaging to be enrolled in the study. Participants will be assigned to one of 7 groups, including cognitively and neurologically normal adults (CN; planned enrollment of n=25); non-amnestic AD (naAD, n=15); frontotemporal lobar degeneration (FTLD) due to tauopathy (FTLD-tau, n=25); FTLD due to TDP-43 (n=12); FTLD-tau due to a known genetic mutation in the MAPT gene (genetic FTLD-tau, n=12); FTLD-TDP due to a known mutation in the GRN gene or open reading frame 72 of chromosome 9 (C9orf72) (genetic FTLD-TDP, n=3); and amnestic MCI/AD (aAD, n=15), Total planned enrollment is thus 107 participants; recruitment and data acquisition for the study are projected to take approximately 6 years.

The current study comprises a baseline visit with a PET/CT imaging scan, using the [18F]-PI-2620 tracer. If funding is available, participants may be asked to return for one or more longitudinal visits to complete a [18F]-PI-2620 brain scan between 12 and 24 months after the previous [18F]-PI-2620 brain scan. These visits must be at least 12 months apart, but ideally not greater than 24 months apart. If a longitudinal visit is missed for any reason, it will not be considered a protocol deviation, and the participant may be scheduled for a [18F]-PI-2620 brain scan as soon as possible thereafter.

The central hypotheses are 1) that [18F]-PI-2620 PET will distinguish Alzheimer's disease (AD) or frontotemporal lobar degeneration (FTLD) tauopathy from the brains of both healthy adults and patients with FTLD due to accumulation of transactive response DNA binding protein 43 kDA (TDP-43); and 2) that in FTLD and AD tauopathies, [18F]-PI-2620 will be associated with patients' current and future cognitive, motor, and functional impairment.

ELIGIBILITY:
Inclusion Criteria: participants must fulfill all of the criteria for one of the following groups.

1. Group 1: cognitively and neurologically normal subjects (CN, n=25)

1. Male or female ≥ 18 years of age currently enrolled in UNICORN (IRB #842873)
2. Cognitively and neurologically normal according to one of the following criteria:

   i. Mini-Mental Status Exam (MMSE; Folstein et al., 1975) score > 27, OR ii. Montreal Cognitive Assessment (MoCA; Carson et al., 2017; Nasreddine et al., 2005) score > 25, OR iii. Global Clinical Dementia Rating of 0, OR iv. Evaluation by a trained clinician
3. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
4. No history of early-onset neurodegenerative disease in biological siblings or parents, based on the investigators' assessment of the participant's self-reported history.

2. Group 2: non-amnestic Alzheimer's disease (naAD, n=15)

1. Male or female ≥ 18 years of age currently enrolled in UNICORN (IRB #842873)
2. Clinically diagnosed by a trained clinician as having a non-amnestic syndrome attributed to likely AD pathology, including but not limited to logopenic-variant primary progressive aphasia (lvPPA), posterior cortical atrophy (PCA), behavioral/dysexecutive AD (bvAD), corticobasal syndrome due to AD (CBS-AD), non-amnestic mild cognitive impairment (naMCI), or non-amnestic AD (naAD).
3. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
4. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.

3. Group 3: FTLD likely due to tau (FTLD-tau, n=25)

1. Male or female ≥ 18 years of age currently enrolled in UNICORN (IRB #842873)
2. Clinically diagnosed by a trained clinician as having a neurodegenerative syndrome likely due to tau , including but not limited to progressive supranuclear palsy (PSP), non-fluent agrammatic primary progressive aphasia (naPPA), corticobasal syndrome (CBS), or behavioral-variant frontotemporal dementia (bvFTD).
3. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
4. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.

4. Group 4: FTLD likely due to TDP-43 (FTLD-TDP, n=12)

1. Male or female ≥ 18 years of age currently enrolled in UNICORN (IRB #842873)
2. Clinically diagnosed by a trained clinician as having a dementia syndrome associated with likely TDP-43 pathology, including but not limited to amyotrophic lateral sclerosis with frontotemporal dementia (ALS-FTD) or semantic-variant primary progressive aphasia (svPPA).
3. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
4. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.
5. Group 5: having a known genetic mutation associated with FTLD-tau (genetic FTLD-tau, n=12)

1. Male or female ≥ 18 years of age 2. Currently enrolled in UNICORN (IRB #842873) with a genetic test result indicating a mutation in the MAPT gene.

3. Clinically diagnosed by a trained clinician as having an appropriate neurodegenerative condition OR confirmed as an asymptomatic mutation carrier.

4. Not clinically depressed, according to one of the following criteria: i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician 5. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.

6. Group 6: having a known genetic mutation associated with FTLD-TDP (genetic FTLD-TDP, n=3)

1. Male or female ≥ 18 years of age
2. Currently enrolled in UNICORN (IRB #842873) with a genetic test result indicating a mutation in the GRN gene or in open reading frame 72 of chromosome 9 (C9orf72).
3. Clinically diagnosed by a trained clinician as having an appropriate neurodegenerative condition OR confirmed as an asymptomatic mutation carrier.
4. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
5. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.

7. Group 7: amnestic Alzheimer's disease (naAD, n=15)

1. Male or female ≥ 18 years of age currently enrolled in UNICORN (IRB #842873)
2. Clinically diagnosed by a trained clinician as having amnestic mild cognitive impairment (MCI) or amnestic Alzheimer's disease (aAD).
3. Not clinically depressed, according to one of the following criteria:

   i. Geriatric Depression scale ≤ 6 (assessed ≤ 6 months prior to study enrollment), OR ii. Evaluation by a trained clinician
4. Have a study partner and LAR (if applicable) who can participate as outlined in the protocol. Please see page 15 for further clarification.

Exclusion Criteria for all groups: Participants will be excluded from enrollment if they meet any of the following criteria.

1. The participant has any medical or psychiatric conditions that, in the opinion of the investigator, would compromise the participant's safety or successful participation in the study.
2. The investigators of UNICORN (IRB #842873) have determined the participant has evidence of structural abnormalities such as major stroke or mass on MRI scan within < 6 months prior to enrollment that is likely to interfere with analysis of the PET scan.
3. The participant is unable to tolerate or have a contraindication to imaging procedures in the opinion of an investigator.
4. Females who are pregnant or breast feeding at the time of the baseline PET/CT scan will not be eligible for this study. A urine pregnancy test will be performed in women of child-bearing potential at screening and within 24 hours of any scheduled PET/CT.
5. The participant has a history of significant past or ongoing alcohol abuse or substance abuse, or dependence based on medical record review or self-reported (may be excluded at the discretion of the investigator.)
6. The participant is enrolled in a clinical trial for a disease-modifying treatment that targets the molecular pathology underlying their neurodegenerative disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Whole brain SUVR | Once during single PET CT
  Whole-brain and regionally specific standardized uptake value ratio (SUVR) calculated over a 30 minute imaging period beginning 45 minutes (groups 1, 2, 4, 6, & 7) after tracer injection
Regional brain SUVR | Once during single PET CT
  Regionally specific standardized uptake value ratio (SUVR) calculated over a 30 minute period beginning at either 30 minutes (groups 3 & 5 plus half of group 1) or 45 minutes (groups 2, 4, & 6 & 7 plus half of group 1) after PET imaging tracer injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Phillips, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advance Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No